CLINICAL TRIAL: NCT00263796
Title: An fMRI Study of the Effect of Intravenous Oxytocin vs. Placebo on Response Inhibition and Face Processing in Autism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anagnostou, Evdokia, M.D. (Individual)
Responsible Party: Principal Investigator, Evdokia Anagnostou, Adjunct Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO # 04-0749 (2)
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitocin (Experimental)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 10 international units = 1 cc, IV over 4 hours
  Other Names: Pitocin
  Arms: Pitocin
Drug: Placebo — Normal Saline, IV over 4 hours
  Arms: Placebo

SUMMARY:
To study the effect of oxytocin on face processing and response inhibition in autistic adults by fMRI.

DETAILED DESCRIPTION:
Autism is a developmental disorder affecting approximately 60/10,000 individuals. It is characterized by social and language deficits and repetitive behaviors/restricted interests. Functional imaging is becoming a very useful tool in trying to understand the neurobiology of autism. Oxytocin is a hormone produced by the brain to assist with labor and lactation. Recent evidence suggests that it may be involved in social attachment and in repetitive behaviors. In this project, we will study how oxytocin changes the way the brain of autistic adults processes faces, and deals with response inhibition (the ability to interrupt ongoing responses should they prove ineffective or interfering with attaining a goal). There is currently no functional imaging data assessing the effect of oxytocin on the brain. We will explore the activation patterns in response to oxytocin across circuits involved in social cognition (face fusiform area) and response inhibition (caudate, orbitofrontal and dorsolateral cortex) by administering a specific fMRI task activating those circuits before and during an oxytocin infusion. We will also explore the effect of oxytocin in these areas by administering specific cognitive testing not associated with fMRI before and during oxytocin infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-IV, ADI, or ADOS criteria for autism spectrum disorder.
2. Age 18-50.
3. Be seen as outpatients
4. IQ>80
5. 5. Demonstrate capacity to provide authorized informed consent or provide consent for participation by an approved surrogate on the autistic individual's behalf

Exclusion Criteria:

1. Subjects who are pregnant or nursing mothers. Sexually active women of childbearing potential who are not using adequate birth control measures.
2. Subjects with epilepsy.
3. Subjects with a history of schizophrenia, schizoaffective disorder or other Axis 1 mental disorders, such as bipolar disorder.
4. Subjects reporting history of encephalitis, phenylketonuria, tuberous sclerosis, fragile X syndrome, anoxia during birth, neurofibromatosis, hypomelanosis, hypothyroidism, Duchenne muscular dystrophy, and maternal rubella
5. Subjects who have received depot neuroleptic medication, or other psychoactive drugs within the past 5 weeks.
6. Subjects with renal or liver disease or abnormalities in blood chemistry.
7. Any metallic prosthesis such as plates, pins and screws, shrapnel, metallic foreign body, vascular or neurosurgical clips that may be incompatible with the MRI and any electrical devices such as a pacemaker or a defibrillator
8. Claustrophobia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2010-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in BOLD with oxytocin infusion | baseline and 4 hours
  Change in BOLD with oxytocin infusion BOLD - blood-oxygen-level-dependent contrast

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States